CLINICAL TRIAL: NCT03084900
Title: Patient-Centered Decision Support to Improve Diabetes Management in Pre-Teens and Adolescents With Type 1 Diabetes
Acronym: CHICAT1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Tamara S. Hannon, Associate Professor, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1612394802; 1DP3DK113183-01 (NIH)
Record Dates: First submitted 2017-03-14; First posted 2017-03-21 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Intervention Arm 1 versus standard care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient-Centered Decision Support (Experimental): Intervention - computer decision support in diabetes clinic. Investigators will use a computerized decision support system to aid clinicians to provide standard of care management while introducing patient-centered guidelines and outcomes measures. The intervention is the use of an electronic decision support tool. The decision support tool consists of a series of questions answered by the patients that will then allow the health care provider to address specific needs during the visit.
  Interventions: Other: Arm 1
- Standard Care (No Intervention): Standard pediatric diabetes care will be compared to the computerized decision support system.

INTERVENTIONS:
Other: Arm 1 — Patient-Centered Decision Support to Improve Diabetes Mgmt. We will use a computerized decision support system to aid clinicians to provide standard of care management while introducing patient-centered guidelines and outcomes measures.The intervention is the use of an electronic decision support tool. The decision support tool consists of a series of questions answered by the patients that will then allow the health care provider to address specific needs during the visit.
  Arms: Patient-Centered Decision Support

SUMMARY:
Investigators propose to study an intervention that will provide patient-centered, automated decision support to diabetes providers with the goals of improving adherence to medical recommendations (both patients and providers), improving self-management, and ultimately improving health outcomes.

DETAILED DESCRIPTION:
Investigators propose to study an intervention that will provide patient-centered, automated decision support to diabetes providers with the goals of improving adherence to medical recommendations (both patients and providers), improving self-management, and ultimately improving health outcomes. Computer decision support systems (CDSS) have scientifically demonstrated advantages for improving care, and the potential to revolutionize diabetes care because they allow for increased reactive and proactive contact with the health care team, real-time adherence support, and intensification of treatment. In this study,investigators will implement the ADA recommended standards of care using a CDSS developed by the research group - the Child Health Improvement through Computer Automation (CHICA) system.9 One of the greatest strengths of the CHICA system is its ability to implement evidence-based recommendations from authoritative sources, in this case the ADA, in a format that integrates easily into routine care. A second strength of the CHICA system is its ability to screen for patient-centered concerns, including barriers to optimal care such as literacy, socioeconomic issues (i.e., food insecurity, housing insecurity, etc.), and mental health issues (i.e., depression). The provider is alerted, and safety mechanisms are set in motion (i.e., referral to mental health provider, etc.) to address identified issues. In order to ensure that we design the most effective CDSS intervention possible, the study team, in collaboration with the Patient Engagement Core (PEC) of the Indiana Clinical and Translational Science Institute, will partner with adolescents, parents, and other stakeholders in a way that exceeds standard expectations for the engagement of these parties in research. Investigators have experience working directly with patients to elucidate patient-centered outcomes, identify determinants of adherence, and to co-design interventions that are inherently more patient-centered.10-14 By combining a patient-centered design approach along with CDSS investigators will be able to individually tailor recommendations to meet the real needs of patients, taking into account the adolescent patient's perspective and input. This truly innovative approach will offer improved technology-based support systems for diabetes management along with attention to patient-centered goals using co-designed interventions for diabetes self-management.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents with type 1 diabetes
2. Parents of adolescents with type 1 diabetes
3. Friends/siblings of adolescents with type 1 diabetes
4. Community partners who work with adolescents with type 1 diabetes
5. Diabetes care providers

   -

   Exclusion Criteria:

   -

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
HbA1c value | 4 years
  Measure of HbA1c value for youth subjects

SECONDARY OUTCOMES:
Hypoglycemia | 4 years
  Number of episodes of hypoglycemia during study
DKA | 4 years
  Number of episodes of DKA during study

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Hannon, MD, Principal Investigator — Indiana University
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No